CLINICAL TRIAL: NCT04264676
Title: Fusobacterium Nucleatum Eradication in Postoperative Stage II/III Colorectal Cancer(FINER-PACE)by Oral Metronidazole: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Clinical Trial.
Brief Title: Study of Oral Metronidazole on Postoperative Chemotherapy in Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Municipal Commission of Health and Family Planning (Other); Ruijin Hospital (Other); Fudan University (Other); Shanghai Zhongshan Hospital (Other); Shanghai Shenkang Hospital Development Center (Unknown)
Responsible Party: Principal Investigator, Jing-yuan Fang, MD, Ph. D, Director of Department of Gastroenterology, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2019-066
Record Dates: First submitted 2020-02-08; First posted 2020-02-11 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Colorectal Cancer Stage II; Colorectal Cancer Stage III
Keywords: Metronidazole; Gut Microbiota; Postoperative Chemotherapy; Colorectal Cancer; Fusobacterium nucleatum
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metronidazole (Active Comparator): supplement of metronidazole 0.4g three times per day for 7 days, which is one treatment every 4 weeks for mFOLFOX6(6 treatments totally),and every 6 weeks for CapeOX (4 treatments totally).
  Interventions: Drug: Metronidazole Oral Tablet
- Placebo (Placebo Comparator): supplement of identical-appearing placebo 0.4g three times per day for 7 days, which is one treatment every 4 weeks for mFOLFOX6 (6 treatments totally),and every 6 weeks for CapeOX 4 treatments totally).
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Metronidazole Oral Tablet — Supplement of metronidazole 0.4g three times per day for 7 days before each two cycles of chemotherapy (mFOLFOX6 once every 4 weeks, CapeOX once every 6 weeks), which is 6 treatments for mFOLFOX6 and 4 treatments for CapeOX totally.
  Arms: Metronidazole
Drug: Placebo oral tablet — Supplement of placebo oral tablet 0.4g three times per day for 7 days before each two cycles of chemotherapy (mFOLFOX6 once every 4 weeks, CapeOX once every 6 weeks), which is 6 treatments for mFOLFOX6 and 4 treatments for CapeOX totally.
  Arms: Placebo

SUMMARY:
Fusobacterium nucleatum (Fusobacterium nucleatum, Fn) has been identified as an independent risk factor for recurrence of colorectal cancer. In this study, oral metronidazole would be used to reduce the abundance of Fn in patients with high Fn, so as to explore whether oral metronidazole can improve the efficacy of postoperative chemotherapy in patients with colorectal cancer.

DETAILED DESCRIPTION:
Gut microbiota are linked to chronic inflammation and carcinogenesis. Chemotherapy failure is the major cause of recurrence and poor prognosis in colorectal cancer patients. Previously in the investigators' research, the investigators find the contribution of gut microbiota to chemoresistance in patients with colorectal cancer. The investigators found that Fusobacterium nucleatum (Fn) was abundant in colorectal cancer tissues in patients with recurrence post chemotherapy, and was associated with patient clinicopathological characterisitcs. Furthermore, the investigators' bioinformatic and functional studies demonstrated that Fn promoted colorectal cancer resistance to chemotherapy. Metronidazole has been known to treat with anaerobe infection, including Fusobacterium. So oral metronidazole would be used to reduce the abundance of Fn in patients with high Fn, so as to explore whether oral metronidazole can improve the efficacy of postoperative chemotherapy in patients with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-75 years
* Individuals firstly confirmed by surgery pathology as colorectal cancer (AJCC cancer staging II - III), who need mFOLFOX6 or CapeOX postoperative chemotherapy
* Individuals with Fn - deltaCT value in colon tissue samples detected by qPCR ≥-12 before receiving chemotherapy
* Individuals who could tolerate chemotherapy drugs: ECOG (Eastern Cooperative Oncology Group) score ≤2 points, WBC(White Blood Cell) ≥4.0×10^9/L, Hb （Hemoglobin） ≥80g/L, PLT （Platelet） ≥80×10^9/L, ALT （Alanine Aminotransferase）< 2ULN （Upper Limmit of Normal）, Scr （Creatinine）< 1.5ULN
* Individuals who participate this study and sign the informed consent form willingly.

Exclusion Criteria:

* Individuals with colorectal adenoma or non-colorectal cancer, such as inflammatory bowel disease
* Individuals with a history of familial adenomatous polyposis (FAP)
* Individuals with severe heart, lung, brain, kidney, gastrointestinal or systemic diseases
* Individuals who used antibiotics for more than 5 days in 1 month prior to chemotherapy
* Individuals with stage I or IV colorectal cancer, or with stage II colorectal cancer who do not need postoperative chemotherapy
* Individuals with contraindications for metronidazole
* Individuals who unwilling to participate this study，or unwilling to sign the informed consent form
* Individuals with any conditions that the researchers considered inappropriate for inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2020-03-31 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival, DFS | 5 years
  The time from the initial surgical treatment of colorectal cancer to the earliest evidence of recurrence.

SECONDARY OUTCOMES:
Overall Survival, OS | 5 years
  The time from the initial surgical treatment of colorectal cancer to death from any cause.
Recurrence Rate, RR | 3 years, 5 years
  Percentage of patients who has recurrence during or after chemotherapy with Metronidazole or Placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Fang, MD, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (4):
- China (4):
  - Division of Gastroenterology and Hepatology, Ren-Ji Hospital, Shanghai Jiao-Tong University School of Medicine, Shanghai Institute of Digestive Disease; Key Laboratory of Gastroenterology & Hepatology, Ministry of Health, Shanghai, Shanghai Municipality
  - Ruijin Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality